CLINICAL TRIAL: NCT04161924
Title: Utilization of Simulated Grid (SimGrid™) Technology for the Reduction of Ionizing Radiation Dose on X-ray Examination in Obese Patients
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Principal Investigator, Roy F Riascos-Castaneda, Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-18-0527
Record Dates: First submitted 2019-11-11; First posted 2019-11-13 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- X-ray imaging with physical grid using conventional processing
  Interventions: Diagnostic Test: X-ray imaging with physical grid using conventional processing
- X-ray without physical grid using conventional processing
  Interventions: Diagnostic Test: X-ray imaging without physical grid using conventional processing
- X-ray imaging without physical grid using experimental SimGrid
  Interventions: Diagnostic Test: X-ray imaging without physical grid using experimental SimGrid offline processing

INTERVENTIONS:
Diagnostic Test: X-ray imaging with physical grid using conventional processing — X-ray imaging with physical grid using conventional processing
  Other Names: GM85
  Groups: X-ray imaging with physical grid using conventional processing
Diagnostic Test: X-ray imaging without physical grid using conventional processing — X-ray imaging without physical grid using conventional processing
  Other Names: GM85
  Groups: X-ray without physical grid using conventional processing
Diagnostic Test: X-ray imaging without physical grid using experimental SimGrid offline processing — X-ray imaging without physical grid using experimental SimGrid offline processing
  Other Names: GM85
  Groups: X-ray imaging without physical grid using experimental SimGrid

SUMMARY:
The purpose of this research study is to learn if a new imaging processing technique called Simulated grid (SimGrid™) will help in getting better quality X-ray images in obese subjects. The GM85 digital radiography machine will be used to obtain X-ray images.

ELIGIBILITY:
Inclusion Criteria:

* Obese adult volunteers with Body-Mass Index (BMI) exceeding 30
* subjects that require at least one X-ray for continuation of care

Exclusion Criteria:

* subject who is known to have lung disease(s) which would interfere with the interpretation of the chest radiography image
* subject who is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients at clinic who needed chest radiography for continuation of care.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Image quality of conventional grid versus SimGrid using 5 point Likert scale | baseline
  Relative image quality will be assessed using a 5 point Likert scale ranging from -2 to +2 with -2 indicating better image quality with conventional grid and +2 indicating better image quality with SimGrid.
Image quality of non-grid versus SimGrid using 5 point Likert scale | baseline
  Relative image quality will be assessed using a 5 point Likert scale ranging from -2 to +2 with -2 indicating better image quality with non-grid and +2 indicating better image quality with SimGrid.

CONTACTS AND LOCATIONS:
Overall Officials: Roy F Riascos-Castaneda, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No